CLINICAL TRIAL: NCT01768169
Title: Phase 2 Study of Metabolic Syndrome Use Omega-3 Fatty Acids and Low Fat Meal Replacements
Brief Title: Study of Metabolic Syndrome Use Omega-3 Fatty Acids and Low Fat Meal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: omega-3 fatty acids
Record Dates: First submitted 2012-12-23; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2012-12

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome,; waist, blood pressure,; fasting plasma glucose,; HDL cholesterol,; triglycerides
MeSH Terms: conditions — Metabolic Syndrome | interventions — Fish Oils

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- fish oil capsule: 10 capsules per day will provide 2130 mg of EPA (1280 mg) and DHA (850 mg)
  Interventions: Dietary Supplement: fish oil capsule

INTERVENTIONS:
Dietary Supplement: fish oil capsule — 500 mg of natural fish oil, made up of 30% omega-3 PUFA (EPA:DHA = 3:2)

SUMMARY:
Increased understanding of the impact of long chain omega-3 PUFAs in combination with a low fat plant-based diet will contribute to decelerating further escalation of the "epidemics" of obesity, the (pre)metabolic syndrome, and T2DM in Taiwan.

DETAILED DESCRIPTION:
The metabolic syndrome is a common condition in which different degrees of hypertension, impaired glucose tolerance, atherogenic dyslipidemia, and central fat accumulation, as well as prothrombotic and proinflammatory states cluster together in the same individual. The modified National Cholesterol Education Program, Adult Treatment Panel III guidelines defined the metabolic syndrome subjects as individuals with 3 or more following criterion:

1. Waist circumference: in male ≥90 cm and female ≥80 cm
2. Raised triglycerides: > 150 mg/dL
3. Reduced HDL cholesterol: <40 mg/dL in males, <50 mg/dL in females
4. Raised blood pressure: systolic blood pressure >130 or diastolic blood pressure >85 mmHg
5. Raised fasting plasma glucose: (FPG)>100 mg/dL

Changes in macronutrient composition have been used to promote weight loss and enhance insulin sensitivity, independent of an emphasis on overall calorie ingestion. Protective effects of fish intake on the development of insulin resistance has been reported in prospective epidemiological studies. Further, long chain omega-3 PUFAs supplementation may improve insulin sensitivity in patients with impaired glucose tolerance and in patients with T2DM.

However, this has not been clearly demonstrated in an intervention trial in Taiwan. Furthermore, the effect of supplementation of long chain omega-3 PUFAs on metabolic risk factors and insulin resistance, except for demonstrated benefit in terms of decreased triglycerides, needs further investigation among Asians.

This 13-week, randomized controlled study will assign approximately 200 subjects meeting criteria for the Metabolic Syndrome (50 each) to the following four arms 1) Standard Taiwan Diet plan; 2) Herbalife meal replacement diet program (Low fat diet); 3) Standard Taiwan Diet plan plus healthy oil supplement (Herbalifeline®) and 4) Herbalife meal replacement plan (Low fat diet) plus healthy oil supplement (Herbalifeline®). All participants will meet with a registered dietitian to assist them with their diet efforts.

In this study, we aim to study the effects of low fat diet with reduced omega-6 PUFAs alone and the same low fat diet with omega-3 fatty acids supplementation on cardiometabolic profile and circulating fatty acid profiles in subjects with the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 65 years
* Female subjects must have a negative pregnancy test at screening, must be surgically sterile or at least 6 months postmenopausal or must use a form of birth control measure.
* BMI of 24 to 40 kg/m2 inclusive.
* Subjects must be in good health other than having metabolic syndrome as determined by medical history, physical examination, and screening clinical laboratory including chemistry panel and CBC.
* Must have stable smoking habits (or be now-smokers) for at least 6 months prior to screening and agree not to intend to change such habits during the course of the study.
* Subjects requiring the regular use of any prescription medication may be admitted to the study providing the dose is stable.
* Ethical subjects only will be admitted who are likely to comply with all visits and instructions. This will be determined in the screening phase.
* Body weight must be stable within 2% of change in the last 3 months.
* Subject must sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or randomization. A subject will be excluded for any condition that might compromise the ability to give truly informed consent for participation in the study.

Exclusion Criteria:

* Diabetes
* nown or documented coronary heart disease (CHD) (including ECG consistent with prior myocardial infraction), cerebrovascular accident (including transient ischemic attack), peripheral vascular disease (including symptoms of claudication)
* Angina or other chest pain that may indicate CHD
* Clinically significant neoplastic, cardiovascular, hepatic, renal, metabolic, endocrine (untreated or unstable), or psychiatric (untreated or unstable)
* Known abnormal liver function tests greater than 3X upper limit of normal
* Smoker, illicit drug use, or excessive alcohol use
* Medications: Lipid lowering therapy, daily NSAID or greater than 325 mg ASA (PRN use ok), clopidogrel (or equivalent), Coumadin, omega-3 fatty acid supplement, other investigational drugs within 30 days of study entry, high omega-3 fatty acid content in diet within past three months
* Pregnancy or planning pregnancy during the study period
* Sensitivity or allergy to fish
* Subjects who had undergone bypass procedure.
* Any debilitating disease such as tuberculosis, HIV etc.
* Unwillingness to give written informed consent for participation in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample, residents of Taiwan
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome index | Day 1 and up to 12 weeks
  1. Waist circumference in male ≥90 cm and female ≥80 cm
  2. Raised triglycerides: > 150 mg/dL
  3. Reduced HDL cholesterol: <40 mg/dL in males, <50 mg/dL in females
  4. Raised blood pressure: systolic blood pressure >130 or diastolic blood pressure >85 mmHg
  5. Raised fasting plasma glucose: (FPG)>100 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yi Huang, Ph.D, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Mecical University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Tang KY, Huang SY, Cheng TM, Bai CH, Chang JS. Haptoglobin phenotype influences the effectiveness of diet-induced weight loss in middle-age abdominally obese women with metabolic abnormalities. Clin Nutr. 2020 Jan;39(1):225-233. doi: 10.1016/j.clnu.2019.01.019. Epub 2019 Jan 26. PMID 30737047